CLINICAL TRIAL: NCT06012019
Title: Characterization of the Immuno-inflammatory Response Involved in Bone Destruction During Periodontitis: Study on Biological Samples With Collection
Brief Title: Periodontitis and Inflammation: Study on Biological Samples
Acronym: CB-PARO2
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230385
Record Dates: First submitted 2023-06-30; First posted 2023-08-25 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-06

CONDITIONS: Periodontitis
Keywords: Periodontitis; Gingivitis; Neutrophils; Subsets; Biological collection
MeSH Terms: conditions — Periodontitis; Gingivitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — gingival tissue and fluid, saliva and serum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Periodontitis Cases: Patients with stage 3 or 4 periodontitis (Chicago 2017) ; BOP ≥ 10%, PD≥ 4mm Patients requiring surgical care such as dental avulsion or pre-prosthetic periodontal surgeries
  Interventions: Other: Biological sampling in Periodontitis Case
- Gingivitis Cases: BOP ≥ 10%, PD≤ 3mm according to Chicago 2017 Patients requiring surgical care such as dental avulsion or pre-prosthetic periodontal surgeries
  Interventions: Other: Biological sampling in Gingivitis Case
- Control: BOP < 10%, PD≤ 3mm Patients with gingival health on intact or reduced periodontium without a history of periodontitis and requiring surgical care such as dental avulsion or aesthetic surgeries
  Interventions: Other: Biological sampling in Control Case

INTERVENTIONS:
Other: Biological sampling in Periodontitis Case — Periodontal bacteria, gingival fluid, unstimulated saliva and blood collection;
  J+7 : tooth extraction : gingival explant sampling
  J+15 : Healing control
  Groups: Periodontitis Cases
Other: Biological sampling in Gingivitis Case — Periodontal bacteria, gingival fluid, unstimulated saliva and blood collection;
  J+7 : tooth extraction or pre-prosthetic periodontal surgeries : gingival explant sampling
  J+15 : Healing control
  Groups: Gingivitis Cases
Other: Biological sampling in Control Case — Periodontal bacteria, gingival fluid, unstimulated saliva and blood collection;
  J+7 : tooth extraction or pre-prosthetic periodontal surgeries : gingival explant sampling
  J+15 : Healing control
  Groups: Control

SUMMARY:
Periodontitis is a major public health problem because it is widespread in the adult population. It leads to the irreversible destruction of the anchoring tissues of the teeth, and represents a modifiable risk factor for systemic inflammatory pathologies. This chronic inflammatory disease, which is associated with oral dysbiosis involving Porphyromonas gingivalis, is triggered by a permissive immune response. It is preceded by a reversible clinical phase, during which there is no bone resorption process: gingivitis. The understanding of the key mechanisms involved in the evolution from gingivitis to periodontitis, which will allow to early identify patient at risk of periodontitis, remain unclear at this time.

Neutrophils are the main cells of inflammation present within the periodontal pockets. The excess of certain neutrophils or the alteration of their functions is associated with the triggering of periodontitis, whereas their activity, finely orchestrated, would be a key to periodontal homeostasis. It is likely that some periodontal bacteria, including P. gingivalis, but also products of matrix catabolism could deregulate the physiological functions of neutrophils towards pro-inflammatory and catabolic profiles. Moreover, to date, the differentiation and role of neutrophil subsets in periodontal homeostasis as well as in gingivitis and its evolution into periodontitis remain poorly studied.

The investigators hypothesize that various subsets of neutrophils may play different roles during the development of periodontitis (evolution of gingivitis to periodontitis).

The primary objective is to characterize neutrophil subtypes associated with periodontal destruction during periodontitis.

Secondary objectives are :

1. Identify specific interactions of tissue-activated neutrophils with the matrix microenvironment during periodontitis
2. Identify specific interactions of tissue or oral (salivary) activated neutrophils with the oral microbiota during periodontitis
3. Identify specific oral (salivary) neutrophil subtypes in periodontal health, gingivitis and periodontitis
4. Evaluate the function, including pro-osteoclastogenic function, of oral neutrophils compared to blood neutrophils stimulated by infection

DETAILED DESCRIPTION:
It's a cross-sectional, monocenter prospective, open-label, non randomized case control study to collect tissue, crevicular, salivary, and serum samples as part of the patient's routine care in oral medicine departments to form a biological collection. The samples and the clinical data of the patients.

Patients will be recruited in the oral medicine departments of AP-HP Charles Foix hospital (Ivry/seine) by periodontists in three groups (Cases : Group 1 : Gingivitis, Group 2 : Periodontitis, and Controls = healthy periodontium. All patients will require surgical care).

The time-line of the research is consistent with the usual patient management in oral medicine departments. Inclusion period is 36 months. There is no specific follow-up due to the research. Gingival tissue sampling during surgery of patients will be performed after their inclusion.

Assessment Criteria :

1. Neutrophil subtypes analysis based on co-expression of neutrophil function markers from a panel of 24 markers by imaging on sections.
2. Identification by immunohistofluorescence (on tissues) of the expression of matrix proteins described as regulating neutrophil function, and search of co-location between these proteins and certain neutrophil subtypes.
3. Identification by immunohistofluorescence (on tissue) of key bacteria of oral dysbiosis in periodontitis, and search for co-localization between these bacteria and certain neutrophil subtypes.
4. Assessment of neutrophil sub-types present in the patient's saliva and study of the correlation within tissue neutrophils during periodontal health, gingivitis and periodontitis.
5. Differentiation and activity of osteoclasts in co-culture with isolated oral /blood neutrophils in patients.

ELIGIBILITY:
Inclusion Criteria:

Common criteria for all patient groups

* Patient > 18 years old
* Patient affiliated to a national health insurance
* Patient who speaks and understands French well enough to be able to read and understand the study information note.
* Patient who does not object to his participation in the study

Specific Criteria :

* Control Group = BOP < 10%, PI<20%, PD≤ 3mm
* Gingivitis cases = BOP ≥ 10%, PD≤ 3mm
* Periodontitis cases = BOP ≥ 10%, PD> 3mm

Exclusion Criteria:

* Patients who have received antibiotic prophylaxis, antibiotic therapy, or anti-inflammatory treatment within 3 months prior to inclusion
* Pregnant or breastfeeding women
* Patients suffering from a disease with defective neutrophil number, activity, activation or function
* Patient deprived of liberty by judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study concerns adult patients consulting the oral medicine department at Hôpital Charles Foix (AP-HP, Ivry sur Seine)
  Cases :
  * Group 1 = Patients should have bacterial gingivitis
  * Group 2 = Patients should have stage 3 or 4 localized or generalized bacterial periodontitis.
  The diagnosis of gingivitis or periodontitis is based on the elements noted during the clinical interview and examination, in accordance with the Chicago 2017 classification.
  Control:
  Patient with healthy gingiva on intact or reduced periodontium with no history of periodontitis, in accordance with the Chicago 2017 classification.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Description of neutrophil subtypes associated with periodontal destruction in periodontitis based on coexpression of markers of neutrophil function . | 36 months
  Distinction of neutrophil subtypes based on coexpression of markers of neutrophil function from a panel of 24 markers by imaging on tissue sections

SECONDARY OUTCOMES:
Identify specific interactions of activated tissue neutrophils with the matrix microenvironment during periodontitis using Immunohistofluorescence identification of the expression of some matrix proteins. | 36 months
  Immunohistofluorescence identification (on tissue) of the expression of matrix proteins described as regulators of neutrophil function, and search for co-localization between said proteins/peptides and certain subtypes of neutrophils
Identify interactions of activated tissue or oral neutrophils with the oral microbiota using Immunohistofluorescence identification of key bacteria and investigation of co-localization between bacteria and certain subtypes of neutrophils | 36 months
  Immunohistofluorescence identification (on tissue) of key bacteria in oral dysbiosis during periodontitis and investigation of co-localization between bacteria and certain subtypes of neutrophils
Describe oral (salivary) neutrophil subtypes during periodontal health, gingivitis and periodontitis based on coexpression of markers of neutrophil function. | 36 months
  Evaluation of neutrophil subtypes present in patient saliva and study of correlation with tissue neutrophils during periodontal health, gingivitis and periodontitis
Evaluate the differenciation, particularly proosteoclastogenic, of oral neutrophils, in comparison with blood neutrophils, stimulated by infection using morphological criteria like the number of nuclei and cell size | 36 months
  osteoclast differentiation will be analyzed using morphological criteria, like the number of nuclei
Evaluate the differenciation, particularly proosteoclastogenic, of oral neutrophils, in comparison with blood neutrophils, stimulated by infection using morphological criteria like the cell size | 36 months
  osteoclast differentiation will be analyzed using morphological criteria, like cell size
Evaluate the activity, particularly proosteoclastogenic, of oral neutrophils, in comparison with blood neutrophils, stimulated by infection, using functional criteria such as resorption activity (size of lacunae formed by the cells on culture dishes) | 36 months
  Osteoclast activity will be assessed by functional criteria such as resorption activity (size of lacunae formed by the cells on specific culture dishes)
Evaluate the activity, particularly proosteoclastogenic, of oral neutrophils, in comparison with blood neutrophils, stimulated by infection, using functional criteria such as expression of activity markers by Trap staining | 36 months
  Osteoclast activity will be assessed by functional criteria such as expression of activity markers (Trap staining)

CONTACTS AND LOCATIONS:
Overall Officials: Marjolaine Gosset, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Charles-Foix Hospital, Ivry-sur-Seine, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal